CLINICAL TRIAL: NCT05137184
Title: A Randomized Controlled, Open-label, Non-inferiority, Three Arm Clinical Study to Assess Inhalation of Low-dose Methoxyflurane, Intranasal Fentanyl, and Intravenous Morphine for Acute Pain in the Pre-hospital Setting
Brief Title: A Comparison of Three Regimens of Acute Pain Management: Methoxyflurane; Intranasal Fentanyl; Intravenous Morphine
Acronym: PreMeFen
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: Sykehuset Innlandet HF (Other); Norwegian Air Ambulance Foundation (Other); University of Oslo (Other)
Responsible Party: Principal Investigator, Fridtjof Heyerdahl, Senior Consultant, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 255159; 2021-000549-42 (EudraCT Number)
Record Dates: First submitted 2021-11-01; First posted 2021-11-30 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Acute Pain; Ambulances
Keywords: Methoxyflurane; Fentanyl; Morphine
MeSH Terms: conditions — Acute Pain | interventions — Methoxyflurane; Fentanyl

STUDY DESIGN:
Masking Description: Masking Statistician
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Methoxyflurane (Experimental): 3 ml inhalation Can be repeated once (3 ml) Maximum total dose of 6 ml
  Interventions: Drug: Methoxyflurane
- Fentanyl IN (Experimental): 100 µg IntraNasal, Patients >70 years: 50 µg IN Can be repeated Maximum total dose 500 µg IN
  Interventions: Drug: Fentanyl
- Morphine IV (Active Comparator): 0.1 mg/kg Intravenous (IV) Patients ≥ 70 years or fragile: 0.05 mg/kg IV Can be repeated Maximum total dose 0.5 mg/kg IV
  Interventions: Drug: Morphine hydrochloride

INTERVENTIONS:
Drug: Methoxyflurane — Inhalation of Methoxyflurane
  Arms: Methoxyflurane
Drug: Fentanyl — Intranasal Fentanyl
  Arms: Fentanyl IN
Drug: Morphine hydrochloride — Intravenous Morphine
  Arms: Morphine IV

SUMMARY:
The study rationale is to provide evidence for early, safe and effective pain management in the ambulance service with non-invasive and fast acting analgesics. Low-dose methoxyflurane and intranasal fentanyl are non-invasive medications that are well-suited for use by ambulance personnel under difficult pre-hospital settings. This is a randomized, controlled, open label, three-arm, non-inferiority, phase 3 drug trial performed in the ambulance service. The randomization will be 1:1:1 to the three treatment groups.

Patients 18 years or older with acute pain with Numeric Rating Scale (NRS) ≥4 with normal physiology and capable of giving informed consent will be included null hypothesis (H0) (tested in hierarchic order a-b-c):

1. Methoxyflurane regimen is inferior to intranasal fentanyl regimen or
2. Methoxyflurane regimen is inferior to IV morphine regimen or
3. Intranasal fentanyl regimen is inferior to IV morphine regimen for treating moderate to severe pain, measured by reduction in Numeric Rating Scale (NRS) 10 minutes after administration.

The study duration for each participant will be from ambulance scene arrival to patient handover in emergency department.

Number of participants: Patient enrolment until successful inclusion of 270 per protocol patients.

Primary endpoint is change in NRS from before administration (t0) to 10 minutes after start of administration (t10).

The study intervention is one of the three IMPs:

* Methoxyflurane: 3 ml inhalation, can be repeated once to a total dose of 6 ml.
* Fentanyl intranasal spray: 100 µg IntraNasal, (patients >70 years 50 µg), can be repeated to maximum total dose 500 µg IN.
* Morphine hydrochloride intravenous: 0.1 mg/kg IV (patients >70 years or fragile 0.05 mg/kg IV), can be repeated to a maximum total dose 0.5 mg/kg IV.

Rescue analgesia is all analgesics other than the allocated IMP. If rescue medication is administered before the assessment of primary endpoint at 10 minutes, the patient will not be part of the per-protocol analysis.

The hypothesis will be tested and the primary endpoint will be evaluated by the 95% confidence limits (95% CI), and a conclusion of non-inferiority will be made if the 95% CI of the estimated treatment difference fully lie within the inferiority margin. Non-inferiority is determined on the basis of a 1-sided equivalence t test on the per protocol population and confirmed, for sensitivity reasons, on the modified intention to treat population.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years of age
2. Acute moderate to severe pain defined by self-reporting pain ≥4 on NRS
3. Capable of giving informed consent
4. Normal physiology

Exclusion Criteria:

1. Life-threatening or limb-threatening condition requiring immediate management
2. Pregnancy or breastfeeding
3. Know allergies, hypersensitivity or serious side effects to opioids or methoxyflurane or other excipients
4. Head injury or medical conditions with neurological impairment (Glasgow Coma Scale (GCS)<14)
5. Previous malignant hyperthermia or persons with suspect genetic predisposition for malignant hyperthermia
6. Massive facial trauma, visible nasal blockage or on-going nose bleeding
7. History of severe liver disease with jaundice and scleral icterus
8. Dialysis or history of severe renal disease (known chronic kidney failure stage 4 or 5)
9. Mono Amine Oxidase-inhibitors last 14 days (pharmacological treatment of depression, Mb Parkinson or narcolepsy)
10. Myasthenia gravis
11. Use of investigational medicinal product (IMP) analgesics 12 hours prior to inclusion
12. Any condition that in the view of the study worker would suggest that the patient is unable to comply with study protocol and procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 338 (Actual)
Dates: Start 2021-11-12 (Actual); Primary Completion 2023-04-22 (Actual); Study Completion 2023-04-22 (Actual)

PRIMARY OUTCOMES:
Change in pain Numeric Rating Scale after 10 minutes | 10 minutes
  Change in Pain Numeric Rating Scale (minimum 0 and maximum 10, higher is worse) from baseline to 10 minutes after start of IMP administration

SECONDARY OUTCOMES:
Change in pain Numeric Rating Scale after 5 minutes | 5 minutes
  Change in Pain Numeric Rating Scale (minimum 0 and maximum 10, higher is worse) from baseline to 5 minutes after start of IMP administration
Change in pain Numeric Rating Scale after 20 minutes | 20 minutes
  Change in Pain Numeric Rating Scale (minimum 0 and maximum 10, higher is worse) from baseline to 20 minutes after start of IMP administration
Change in pain Numeric Rating Scale after 30 minutes | 30 minutes
  Change in Pain Numeric Rating Scale (minimum 0 and maximum 10, higher is worse) from baseline to 30 minutes after start of IMP administration
Need for rescue analgesia | 2 hours
  Number of patients with administration of rescue analgesia
Type of rescue analgesia | 2 hours
  Type of rescue analgesia administered
Dose of rescue analgesia | 2 hours
  Dose of rescue analgesia administered
Route of administration of rescue analgesia | 2 hours
  Route of administration of rescue analgesia
Time from ambulance arrival to IMP administration | 1 hour
  Time from arrival of ambulance personnel by the patient to administration of IMP
Time from ambulance arrival to 2-point NRS reduction | 1 hour
  Time from ambulance arrival to first measure of a reduction in NRS of 2 points or more
Change in level of sedation | 30 minutes
  Change in GCS from baseline to 10 and 30 minutes
Change in respiration | 30 minutes
  Change in respiratory rate from baseline to 10 and 30 minutes
Change in blood pressure | 30 minutes
  Change in systolic blood pressure from baseline to 10 and 30 minutes
Health Care Personnel Likert Scale | 2 hours
  Likert Scale (1 to 5, higher is better) of health care professional satisfaction at end of mission
Patient Likert Scale | 2 hours
  Likert Scale (1 to 5, higher is better) of patient satisfaction at end of mission
Numbers of patients with adverse events in each treatment group | 2 hours
  Registration of adverse events during study period until end of intervention and compare numbers of patient with adverse events in each group

OTHER OUTCOMES:
Change in pain Numeric Rating Scale after 10 minutes stratified by diagnosis groups | 30 minutes
  Change in Pain Numeric Rating Scale (minimum 0 and maximum 10, higher is worse) stratified by diagnosis groups
Need for rescue medication related to painful procedures | 2 hours
  Proportion of patient receiving rescue treatment related to procedures (reposition of fractures, relocation etc)
Number of vascular cannulation attempts in each patient | 2 hours
  Attempts and success of vascular cannulation access in each patient, stratified by treatment allocation
Ambulance worker competence influence on change pain Numeric Rating Scale after 10 minutes | 2 hours
  Change in Pain Numeric Rating Scale (minimum 0 and maximum 10, higher is worse) from baseline to 10 minutes after start of IMP administration stratified by ambulance worker competence (educational levels)
Ambulance worker competence influence on patient satisfaction Likert Scale | 2 hours
  Likert Scale (1 to 5, higher is better) of patient satisfaction at end of mission, stratified by ambulance worker competence (educational levels)
Change in pain Numeric Rating Scale after 10 minutes in acute coronary syndrome patients | 2 hours
  Change in Pain Numeric Rating Scale (minimum 0 and maximum 10, higher is worse) from baseline to 10 minutes after start of IMP administration stratified by the presence of acute coronary syndrome defined by troponin elevation higher than 99 percentile or significant ST-segment elevation on any ECG lead.

CONTACTS AND LOCATIONS:
Overall Officials: Fridtjof Heyerdahl, MD PhD, Principal Investigator — Senior Consultant
Locations (1):
- Sykehuset Innlandet, Gjøvik, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Simensen R, Fjose LO, Thorsen K, Olsen IC, Rehn M, Hagemo J, Smalberget L, Heyerdahl F. Comparison of inhalational methoxyflurane, intranasal fentanyl, and intravenous morphine for treatment of prehospital acute pain in Norway (PreMeFen): a randomised, non-inferiority, three-arm, phase 3 trial. Lancet. 2026 Dec 20;406(10522):2957-2967. doi: 10.1016/S0140-6736(25)01575-2. Epub 2025 Nov 20. PMID 41275876